CLINICAL TRIAL: NCT05312957
Title: Evaluation of the Analgesic Effect of Erector Spinae Plane Block in Patients Undergoing Coronary Artery Bypass Graft Surgery: A Randomized Controlled Trial Study
Brief Title: Efficacy of Erector Spinae Plane Block in Caridac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AbantIBU mb6
Record Dates: First submitted 2021-12-15; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Pain
Keywords: Erector spinae plane block,; coronary artery bypass graft surgery,; postoperative pain.; opioid consumption
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Group ESP;The probe was placed craniocaudally in the parasagittal plane approximately 3 cm lateral to the T5 spinous process T5 transverse process is detected. When the block needle (Stimuplex B. Braun R, Melsungen, Germany) touched the transverse process, 0.5-1 mL of the 0.9% NaCl test dose was administered between the erector spinae muscle fascia and the vertebral transverse process, and the needle location was confirmed. Then, 20 ml of 0.25% bupivacaine was administered to this area, and an ESP block was applied Group Control : no intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ESP (Active Comparator): The probe was placed craniocaudally in the parasagittal plane approximately 3 cm lateral to the T5 spinous process. The T5 transverse process is detected and When the block needle touched the transverse process,Then, 20 ml of 0.25% bupivacaine was administered to this area, and an ESP block was applied
  Interventions: Other: erector spinae plane block
- Group Control (No Intervention): Group Control: Tramadol HCL was administered from vein with a patient-controlled analgesia device after extubation.

INTERVENTIONS:
Other: erector spinae plane block — Group ESP (Arm 1)The probe was placed craniocaudally in the parasagittal plane approximately 3 cm lateral to the T5 spinous process. The T5 transverse process is detected .When the block needle (Stimuplex B. Braun R, Melsungen, Germany) touched the transverse process, 0.5-1 mL of the 0.9% NaCl test dose was administered between the erector spinae muscle fascia and the vertebral transverse process, and the needle location was confirmed.Then, 20 ml of 0.25% bupivacaine was administered to this area, Group Control (Arm 2) :No intervention
  Arms: Group ESP

SUMMARY:
Introduction: Opioid-based pharmacological treatment is frequently used in the treatment of pain after coronary artery bypass graft (CABG) surgery. If adequate postoperative analgesia is not provided in such surgeries, pulmonary and cardiovascular complications may develop. This study aimed to provide effective analgesia and reduce postoperative opioid consumption by applying preemptive erector spinae plane (ESP) block.

Methods: A total of 50 patients who underwent CABG surgery were included in this prospective randomized controlled study. Patients were randomly divided into two groups: the ESP group and the control group. The intervention to the ESP group was applied bilaterally at the T5 level before the surgery. The primary outcome was postoperative opioid consumption; the other outcomes included visual analog scale scores, intraoperative opioid consumption, and duration of hospital stay.

DETAILED DESCRIPTION:
Study Design and Patient: This prospective randomized study was conducted with the approval of the local ethics committee of the Bolu Abant Izzet Baysal University in Turkey (Approval date 03/11/2020; Decision no. 2020/243). All patients who agreed to participate in the study were informed about the purpose of the study and the anesthesia method to be used, and their written consent was obtained. Sixty-five patients, aged 50-75 years, at the risk of American Society of Anesthesiologists (ASA) III, who was planned off-pump CABG surgery were invited to the study between November 2020 and April 2021. In the preoperative evaluation, patients with hypersensitivity to the drugs to be used or the substances in their composition, having moderate or severe left ventricular dysfunction, bleeding disorders, liver and kidney failure, chronic obstructive pulmonary disease, patients who do not have sufficient intellectual capacity to use the PCA device, and who refused to participate in the study were excluded from the study. In the intraoperative period, patients who needed a cardiopulmonary bypass pump and those who needed an aortic balloon pump support were excluded from the study. In the postoperative period, patients for whom the extubation duration was longer than four hours and those who required re-exploration were excluded from the study The groups were randomized; It was divided into Group E (ESP Group) and Group C (Control Group). The Ramdom.org program (https://www.random.org/lists/?mode=advanced) was used for the randomization of the groups. Demographic data (gender, age, weight, height, body mass index (BMI)) of all patients were recorded. The patients were taken to the operating room without premedication. and electrocardiography (ECG), heart rate (HR) Sist, and peripheral oxygen saturation (SpO2) values were monitored and two peripheral vascular accesses were established with an 18-gauge intravenous (IV) cannula. To provide continuous arterial blood pressure monitoring, the radial artery was cannulated by applying topical anesthesia after the Allen test.

Interventions In Group E patients, a prone position was given before general anesthesia induction. Compliance with the rules of asepsis-antisepsis was achieved. A Sonosite-180 Plus model USG (L38/10-5 MHz Transducer, SonoSite Inc., Bothell, WA 98021 USA) was used for the intervention. An adjusted linear probe was used, which was set to a depth of 2-5 cm and a frequency of 10-15 MHz. The probe was placed craniocaudally in the parasagittal plane approximately 3 cm lateral to the T5 spinous process. The T5 transverse process is detected using a planal approach. Before the procedure, the skin, subcutaneous tissue, trapezius, rhomboid, and erector spinae muscles were identified, and local anesthesia was administered using 2% lidocaine (Aritmal 2% ampoule, Osel Medicine Istanbul, Turkey). When the block needle (Stimuplex B. Braun R, Melsungen, Germany) touched the transverse process, 0.5-1 mL of the 0.9% NaCl test dose was administered between the erector spinae muscle fascia and the vertebral transverse process, and the needle location was confirmed. Then, 20 ml of 0.25% bupivacaine (Buvasin 0.5% Vem Medicine Istanbul, Turkey) was administered to this area, and an ESP block was applied (Figure 1). The same procedure was performed on the opposite side, and a bilateral ESP block was applied. The block was considered successful when cold loss developed. No preoperative procedure was applied to the Group C patients.

Anesthetic Management For the induction of general anesthesia, 2 µg/kg fentanyl (Talinat 50 mcg/ml VEM İlaç San. ve Tic. A.Ş. İstanbul, Turkey), 2 mg/kg propofol (Propofol Lipuro 1% 10mg/ml ampoule, B. Braun, Melsungen, Germany), and 0.6 mg/kg rocuronium (Esmeron 50mg/5ml Merck Sharp Dohme İlaçları Ltd. Şti. Levent/Istanbul) were given intravenously and the patient was intubated after adequate muscle relaxation was achieved. Then, central venous access was achieved. For anesthesia maintenance, 2% sevoflurane (Sevorane® Liquid 100%, AbbVie, Queenborough Kent, England) was used in 50% air and 50% oxygen. Fentanyl (0.5-2 mcg/kg) was administered 1-2 minutes before the thorax incision. An additional 1-2 mcg/kg of intravenous (IV) fentanyl was administered to patients with a 20% increase in blood pressure or heart rate. After induction, 1 mcg/kg fentanyl, and 0.25 mg/kg rocuronium were administered at half-hour intervals in both groups. Before cross-clamping the ascending aorta, the systolic pressure had aimed to be below 100 mmHg. To maintain a systolic pressure below 100 mmHg, patients were administered 1-2 mcg/kg fentanyl when necessary. Intraoperative fentanyl consumption was recorded. During anesthesia, intermittent arterial blood gas monitoring was performed on all patients. The anesthesia and surgery durations of the patients were recorded, and they were taken to the intensive care unit (ICU) as intubated after the operation. The patients were extubated within 4 hours postoperatively. Patient-controlled analgesia devices were applied to all patients after extubation. Tramadol HCl (Tramosel 100 mg/2 ml Haver Pharma İlaç A.Ş, Istanbul/Turkey) was adjusted as IV bolus 20 mg doses of tramadol HCl every time a button was pressed, at a concentration of 5mg/ml. The device was adjusted to allow a maximum dose of 400 mg in 24 hours, with a lock-in time of 20 minutes; total tramadol consumption was recorded. After extubation, VAS values were recorded at the 1st, 2nd, 4th, 8th, 12th, 18th, 24th, 36th, and 48th postoperative hours. During the 0-1, 1-12, 12-24, 24-36, and 36-48 time zones, heart rate, systolic blood pressure, mean blood pressure, diastolic blood pressure, and peripheral oxygen saturation were monitored and recorded. Nausea, vomiting, pruritus, desaturation, urinary retention, and other side effects were followed up and recorded in the patient follow-up after extubation. Postoperative nausea and vomiting were treated with 4mg of ondansetron (IV) (Ondaren 4mg/2ml Vem İlaç A.Ş Istanbul, Turkey), and rash and itching with 45.5 mg of pheniramine (IV) (Avil amp 45.5mg/2ml Sandoz İlaç A.Ş. Istanbul/Turkey). When the VAS was above four, IV 0.05 mg/kg morphine (Morphine HCL® 0.01 g/ml amp Galen İlaç A.Ş./Turkey) was administered as rescue analgesia. The extubation and ICU discharge times of the patients in both groups were recorded

ELIGIBILITY:
Inclusion Criteria:

* aged 50-75 years,
* at the risk of American Society of Anesthesiologists (ASA) III,
* patients who were planned off- pump CABG surgery

Exclusion Criteria:

* In the preoperative evaluation,

  * patients with hypersensitivity to the drugs to be used or the substances in their composition
  * patients moderate or severe left ventricular dysfunction, with bleeding disorders, with liver and kidney failure, with chronic obstructive pulmonary disease
  * patients who do not have sufficient intellectual capacity to use the PCA device,
  * patients who refused to participate in the study ----In the intraoperative period, patients who needed a cardiopulmonary bypass pump and those who needed an aortic balloon pump support -----In the postoperative period, patients for whom the extubation duration was longer than four hours and those who required re-exploration were excluded from the study

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
measuring opioid consumption after surgery | 0-1hours
  tramadol consumption (mg)
measuring opioid consumption after surgery | 1-12hours,
  tramadol consumption (mg)
measuring opioid consumption after surgery | 12-24hours,
  tramadol consumption (mg)
measuring opioid consumption after surgery | 24-36hours,
  tramadol consumption (mg)
measuring opioid consumption after surgery | 36-48hours
  tramadol consumption (mg)

SECONDARY OUTCOMES:
Evaluation of the postoperative visual analog scale(VAS) score | 1st hours
  postoperative VAS score ( VAS ;subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain.")
Evaluation of the postoperative VAS score | 2nd hours
  postoperative VAS score(0 no pain-10 "worst pain.")
Evaluation of the postoperative VAS score | 4th hours
  postoperative VAS (0 no pain-10 "worst pain.")
Evaluation of the postoperative VAS score | 8th hours
  postoperative VAS score (0 no pain-10 "worst pain.")
Evaluation of the postoperative VAS score | 12th hours
  postoperative VAS score (0 no pain-10 "worst pain.")
Evaluation of the postoperative VAS score | 18th hours
  postoperative VAS score (0 no pain-10 "worst pain.")
Evaluation of the postoperative VAS score | 24thhours
  postoperative VAS score (0 no pain-10 "worst pain.")
valuation of the postoperative VAS score | 36th hours
  postoperative VAS score (0 no pain-10 "worst pain.")
valuation of the postoperative VAS score | 48th hours
  postoperative VAS score (0 no pain-10 "worst pain.")

CONTACTS AND LOCATIONS:
Locations (1):
- Abant Izzet Baysal University Medical School,, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No